CLINICAL TRIAL: NCT03020173
Title: The Difference Seen in Granulosa Cells and Immature Oocytes in IVF Treated Patients Sorted by Body Mass Index (BMI)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0098-16
Record Dates: First submitted 2017-01-02; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BMI above 30: Oocytes and granulosa of infertile women with BMI above 30
  Interventions: Other: Laboratory study
- BMI below 30: Oocytes and granulosa of infertile women with BMI above 30
  Interventions: Other: Laboratory study

INTERVENTIONS:
Other: Laboratory study — Laboratory analysis to determine composition of granulosa and oocytes

SUMMARY:
This study aims to discover the connection between BMI and oocyte and granulosa consistencies.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women undergoing IVF
* Consent to participate in study

Exclusion Criteria:

* Fertility preservation due to cancer
* Endocrine disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing IVF treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of composition of granulosa cells and oocytes | One year
  Laboratory measurement of lipid and cholesterol amounts, mitochondrial distribution and telomere length according to BMI levels

IPD SHARING:
Plan to Share IPD: No